CLINICAL TRIAL: NCT05807594
Title: Efficacy of a Novel Digital Platform to Scale-Up a Personalized Prenatal Weight Gain Intervention Using Control Systems Methodology
Brief Title: Healthy Mom Zone Gestational Weight Gain Management Intervention 2.0
Acronym: HMZ Two
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Principal Investigator, Danielle Downs, Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00019075
Record Dates: First submitted 2023-03-06; First posted 2023-04-11 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Gestational Weight Gain; Overweight and Obesity; Pregnancy; Energy Balance
MeSH Terms: conditions — Gestational Weight Gain; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: A staff member will request randomization after the pre-intervention measures by unique subject ID number. The study biostatistician will develop the randomization scheme using variable-size, random permuted blocks to ensure the number of subjects in each group is balanced after each set of B randomized subjects where B is block size. Randomization to control (n=72) and intervention (n=72) groups will use 1:1 allocation; subjects will be entered consecutively. Randomization will be stratified by pre-pregnancy BMI status (< 29.9 kg/m2 vs. greater than or equal to 30 kg/m2). A staff member will call each woman to inform her of study assignment and schedule her for the first session (attention control or HMZ 2.0 intervention).
Masking Description: All investigators and the outcomes assessor(s) will be masked from the randomization scheme, and what study groups each participant will be/was randomized to. The randomization scheme will be developed and programmed into REDCap by the biostatistician. The team of investigators will not have knowledge of the randomization scheme or be able to view the programming. The programming will be password protected and only be able to be accessed by the biostatistician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HMZ 2.0 Intervention Group (Experimental): HMZ 2.0 will be delivered by a registered dietitian in weekly didactic, one-on-one discussions in remote synchronous format (e.g., Zoom). If a subject has internet connectivity issues, she will be able to participate in the remote sessions from an onsite location (e.g., laboratory space on the Penn State University Park campus, clinical space at Hershey campus or Geisinger). All intervention women will receive the baseline intervention delivered as a maximum of 24 weekly modules (depending on gestational age at enrollment) which includes: Education and Counseling (GWG/PA/EI/sedentary behaviors/sleep behaviors/stress management, etc.), Goal-Setting and Action Plans (guided and self-selected PA/EI goals including recipe and workout booklet use), Self-Monitoring (wearing/using mHealth tools to monitor GWG/PA/EI/sleep), and Featured Evidence and Fetal Growth Facts (evidence-based studies and baby growth fun facts shared with women about how mom's health impacts her baby).
  Interventions: Behavioral: HMZ 2.0 Intervention
- Attention Control Group (Active Comparator): All women will receive prenatal care offered by recruitment sites with routine provider visits, prenatal counseling, brief discussions on healthy prenatal behaviors, and clinical oversight of health (e.g., monitor glucose levels if diagnosed with gestational diabetes during the study period). Women randomized to the attention control group will complete the same measurement procedures as the intervention group. To match the HMZ intervention group, women will receive weekly, remote-delivered education content (60 min/session) on preparing for labor/delivery and benefits of behavioral pain management strategies (e.g., mindfulness-based relaxation, imagery, music, massage, deep-breathing) to regulate pain after childbirth with non-pharmacological approaches. Content is drawn from evidence-based guidelines and materials designed by Dr. Downs and her team for a Patient-Provider Toolbox to reduce opioid-related pain management use after childbirth.
  Interventions: Behavioral: Attention Control Intervention

INTERVENTIONS:
Behavioral: HMZ 2.0 Intervention — The intervention may be adapted such that a woman receives more support with each adaptation (only women who need added support to regulate GWG will receive adaptation). The model-based predictive control system in the HMZ 2.0 digital platform will continually and automatically evaluate GWG, identify when a woman may exceed GWG guidelines, and recommend an adaptation. The registered dietitian will review the data and behavior strategies that are suggested (guided PA workouts, EI cooking demonstrations, customized grocery planning, portion size control, food scales, and meal replacements). Practical, easy-to-adopt examples will be provided (walking in 5-10 min increments throughout the day to increase PA kcal, reduce sitting by 5 min/hour; replace 8 oz of whole milk with skim milk to reduce EI kcal) to facilitate behavior change while adhering to safety standards. Each woman's unique preferences and past successes with strategies are also considered when personalizing the dosage.
  Arms: HMZ 2.0 Intervention Group
Behavioral: Attention Control Intervention — Consistent with guidelines for comparator groups, all women will receive prenatal care offered by recruitment sites with routine provider visits, counseling about prenatal behaviors (e.g., no smoking), and clinical oversight of health. Women randomized to the attention control group will complete the same measurement procedures as the intervention group.
  Arms: Attention Control Group

SUMMARY:
The goal of this clinical trial is to see if the enhanced HMZ 2.0 intervention with new control system/digital platform to regulate gestational weight gain (GWG) and impact maternal-infant outcomes while collecting implementation data works and can be given to other pregnant women in various settings. The question this study aims to answer are:

1. Does the new intervention manage GWG?
2. Does the new intervention have any influence on sleep and eating behaviors and infant outcomes.
3. Does the new platform and other data collected help inform how well the research and information can be used in health care settings?

144 pregnant women with overweight/obesity will be randomized to either the HMZ 2.0 intervention or attention control groups from ~8-36 weeks gestation. All participants will be asked to:

1. Weight themselves and wear an activity monitor each day over the study.
2. Complete online surveys at either a weekly or monthly level about their thoughts, attitudes, and behaviors on GWG, physical activity, eating behaviors, sleep, their anxiety, depression, and stress.
3. Attend weekly sessions with a registered dietician.

The weekly sessions will differ based on intervention group. The HMZ 2.0 intervention group will receive education, create and follow goal-setting and action plans, self-monitor their behaviors, and receive feature evidence and fetal growth facts. Education, goals, and self-monitoring will focus on GWG, physical activity, eating behaviors, sleep, self-regulating behaviors and emotions, and preparing for labor/delivery and postpartum.

The attention control group will receive weekly sessions on preparing for labor/delivery and benefits of behavioral pain management strategies (e.g., mindfulness-based relaxation, imagery, music, massage, deep-breathing) to help with pain after childbirth without medicine.

DETAILED DESCRIPTION:
Pre-intervention: Onsite procedures. Pregnant women with overweight/obesity enrolled in the study will be asked to complete assessments (≥8 and <18 weeks gestation) at the Penn State Clinical Research Center (University Park or Hershey campus) or at home via Zoom. A study staff member will describe the study and obtain consent. Women with any health issues will be asked to follow-up with their provider and/or given a referral as needed. Subjects will have access to REDCap (Research Electronic Data Capture), a secure, web-based application to complete online surveys for social cognitive outcomes for PA and EI (eating healthy/ limiting unhealthy foods), and sleep and eating behaviors. A staff member will answer questions and explain the free-living procedures. This visit will take ~90 minutes.

Pre-intervention: Free-living procedures. A 7-9-day period will provide a grounding of each subject's baseline physical activity (including sedentary behavior), energy intake, social cognitive determinants, and sleep/eating behaviors for the individual energy balance model to predict GWG. Energy intake kcal will be estimated with the back-calculation method utilizing measured weight, physical activity, and resting metabolic rate (quadratic regression formula). There is not a set threshold of data compliance for back-calculating energy intake, the investigators will use strategies to reach similar compliance (>90%) as our feasibility trial and other studies that used a run-in phase. Only women with no weight or physical activity data during this period will be excluded. On the morning of each day of the 7-9-day free-living protocol, subjects will be asked to complete study measures. The investigators will prompt with daily reminders and follow-up with non-compliant women to resolve barriers/technology issues.

Measurement procedures over study period. Subjects will use mHealth tools for real-time data collection on our energy balance and behavior model constructs to predict GWG in the Control Optimization Trial and assess sleep/eating behaviors. Data collection will occur: daily for GWG and physical activity/sedentary behavior/sleep; weekly for physical activity/energy intake social cognitive determinants (online in REDCap), and on at least 2 weekdays/1 weekend for energy intake diet quality. Monthly measures of eating behaviors and psychosocial health will be assessed.

Post-intervention assessments. Maternal GWG, physical activity, sedentary behavior, energy intake, social cognitive determinants, and sleep/eating behaviors will be obtained with the same mHealth devices/procedures as described above in the pre-intervention assessments. To reduce subject burden, there will be no onsite post-assessments.

Labor and delivery data will be abstracted from the medical record with patient HIPAA authorization.

Randomization. A staff member will request randomization after the pre-intervention measures by unique subject ID number. The study biostatistician, will develop the randomization scheme using variable-size, random permuted blocks to ensure number of subjects in each group is balanced after each set of B randomized subjects where B is block size. Randomization to control (n=72) and intervention (n=72) groups will use 1:1 allocation; subjects will be entered consecutively. Randomization will be stratified by pre-pregnancy BMI status (< 29.9 kg/m2 vs. ≥ 30 kg/m2). A staff member will call each woman to inform her of study assignment and schedule her for the first session (attention control or HMZ 2.0 intervention).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* ≥ 8 and < 18 weeks gestation at time of screening. This range of gestational age is chosen to: a) reduce chances of false pregnancy or miscarriage under 8 weeks gestation and b) recruit women in the 1st trimester for greatest impact of the intervention on gestational weight gain. In the feasibility and initial impact study, the investigators had less than 10% (n=3) miscarriages prior to randomization using these criteria
* Singleton gestation
* Not currently heavily smoking (>20 cigarettes/day)
* Any parity (i.e., first-time pregnancy, second pregnancy, etc.)
* Any race/ethnicity
* Ages 18-45 years
* Body mass index (BMI) range 20.0 to 45.0. If BMI is over 40, consultation with woman's health care provider will be made to determine eligibility and ensure she does not have any contraindications to physical activity or other concerns with intervention participation.
* Haven't exceeded 25% or more of their total GWG (based on BMI and IOM guidelines) from pre-pregnancy to date of enrollment.
* Participant has physician consent to confirm subject participation
* Able to read, understand, and speak English
* Access to a computer/phone
* Willingness and ability to complete study materials and intervention sessions electronically (e.g., email, Facetime, Zoom), at home (e.g., Zoom sessions delivered synchronous and asynchronous) or if requested by the participant, on-site at Penn State University Park or Hershey campuses.
* No current use of weight loss medications
* No current participation in another interventional study or program that influences weight control
* No planned bariatric surgery during this current pregnancy
* No absolute contraindications to exercise in pregnancy and relative contraindications with provider consent (see below)

Exclusion Criteria:

* Not pregnant women
* Men (unable to become pregnant)
* Multiple gestation
* < 8 weeks gestation or > 18 weeks gestation at time of pre-intervention assessment
* Currently smoking > 20 cigarettes/day
* Outside of the age range of 18-45 years
* Outside of the BMI range of 20.0-45.0
* Exceeded 25% of their total GWG (based on BMI and IOM guidelines) from pre-pregnancy to date of enrollment
* Not able to read and/or understand English
* Unable to access materials by computer or phone (even with data plan assistance if necessary)
* Current use of weight loss medications
* Current participation in another interventional study or program that influences weight control
* Planned bariatric surgery during this current pregnancy
* Contraindications to aerobic exercise in pregnancy:

Absolute contraindications to exercise:

* Hemodynamically significant heart disease
* Restrictive lung disease (pulmonary fibrosis, sarcoidosis, pleural effusion, neuromuscular disease). This DOES NOT include ASTHMA
* Incompetent cervix/cerclage
* Severe anemia
* Multiple gestation at risk for premature labor
* Persistent 2nd or 3rd trimester bleeding
* Placenta previa after 26 weeks gestation
* Premature labor during the current pregnancy
* Ruptured membranes
* Poorly controlled chronic hypertension
* Preeclampsia diagnosis during current pregnancy
* Poorly controlled Type 1 diabetes

Relative contraindications to exercise (if permission is not given by provider):

* Unevaluated maternal cardiac arrhythmia
* Chronic bronchitis
* Extreme morbid obesity (BMI > 40.0; needs provider consent to participate)
* Extreme underweight (BMI < 12.0)
* History of extremely sedentary lifestyle
* Current eating disorder(s) diagnosis
* Severe food allergies and/or dietary restrictions that may preclude study participation.
* Intrauterine growth restriction in current pregnancy
* Poorly controlled respiratory disorder (severe asthma) that precludes study participation
* Orthopedic limitations
* Poorly controlled seizure disorder
* Poorly controlled thyroid disease
* Uncontrolled sleep disorder (insomnia, sleep-disordered breathing)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Gestational Weight Gain and Weight Change | Measured daily at pre-post intervention and daily throughout the intervention study period (~6 months).
  Weight and GWG will be assessed daily at home using the FitBit Aria Air Smart Scale (weights will be uploaded to online program via Bluetooth). GWG will be standardized: target weight gain will be determined for each woman based on BMI status (OW = 15-25 lb., OB = 11-20 lb.). For the criterion measure to determine when to adapt the intervention, weight gain will be calculated to determine if a woman is gaining < her goal (-), at the exact amount of her goal (0), or > her goal (+). Pre-pregnancy weight and GWG from the first prenatal visit to the last pre-delivery weight will also be obtained from clinical records. Weight will also be assessed at the Penn State Clinical Research Center using standard procedures (measured in duplicate to nearest kg using a high precision stand-on adult scale).
Physical Activity (PA) and Sedentary Behavior | Measured daily at pre-post intervention (Fitbit Charge 5 and ActiGraph) and daily (Fitbit Charge 5) throughout the intervention study period (~6 months).
  Women will wear the wrist-worn Fitbit Charge 5 (Fitbit Inc., San Francisco, CA) 24 hours/day from the pre-intervention assessment until the end of the post-intervention assessment. The Fitbit Charge 5 will be used for continuous PA measure for our energy balance model to predict GWG. It will measure activity kcal, steps, minutes in sedentary/light/moderate PA. The waist-mounted ActiGraph GT3X will be worn at pre- and post-intervention during waking hours to assess PA and sedentary behavior (activity kcal, steps, minutes in sedentary/light/moderate PA). While the ActiGraph is considered a "gold standard" PA measure, our pilot data showed high burden for PW-OW/OB to wear it continuously; thus, it will be used as a pre-post intervention PA measure only.
Energy Intake (EI) Estimation (Back-Calculation of Energy Intake) | Measured at pre-post intervention and daily throughout the intervention study period (~6 months).
  Self-report EI measures under-estimate EI by 35-59%; EI under-reporting is common in people with obesity and especially in PW-OW/OB. Because our energy balance model relies on accurate EI/PA estimates to predict GWG (and our PA/weight measures provide accurate estimates), EI under-reporting compromises the prediction. EI is estimated from measured W (Aria Wi-Fi scale), PA (Fitbit Charge 5 activity monitor), and resting metabolic rate (RMR; Breezing mobile metabolism device) with k=1, 2,… N relating to day 1- day N. T is the sampling time (T=1 day). The noise in W is small relative to the total W, but the extent of this noise can affect the calculated rate of GWG/day, so a 5-day moving average filter is used to preprocess (smooth) measured W before "true" daily EI is estimated.

SECONDARY OUTCOMES:
Theory of Planned Behavior Constructs: Healthy Eating/Limit Unhealthy Eating Attitude, Subjective Norm, Perceived Behavioral Control, Intention | Measured at pre-post intervention, daily during the 10-day free-living period, and weekly throughout the intervention study period (~6 months).
  The Theory of Planned Behavior will inform our dynamical model in order to create individualized interventions for OW/OBPW. Beliefs: These items were developed to assess Theory of Planned Behavior (TPB) behavioral, control, and normative beliefs. Main Constructs: The Theory of Planned Behavior (TPB) Healthy Eating Main Constructs measure is a 38-item measure developed to assess the main constructs of the TPB (i.e., attitude, subjective norm (SN), perceived behavioral control (PBC), intention) as they relate tohealthy eating behavior. Scoring for the TPB is the sum of each subscale. Attitude and Limit Attitude range of scores: 7-49 - higher score means greater/more positive attitude; SN and Limit SN range: 3-21 - higher score greater/more positive subjective norm; PBC and Limit PBC range: 3-21 - higher score greater/more positive PBC; Intention range: 6-42 - higher score greater/more positive intention.
Theory of Planned Behavior Constructs: Physical Activity Attitude, Subjective Norm, Perceived Behavioral Control, Intention | Measured at pre-post intervention, daily during the 10-day free-living period, and weekly throughout the intervention study period (~6 months).
  The Theory of Planned Behavior will inform our dynamical model in order to create individualized interventions for OW/OBPW. Beliefs: These items were developed to assess Theory of Planned Behavior (TPB) behavioral, control, and normative beliefs. Main Constructs: The Theory of Planned Behavior (TPB) Healthy Eating Main Constructs measure is a 38-item measure developed to assess the main constructs of the TPB (i.e., attitude, subjective norm (SN), perceived behavioral control (PBC), intention) as they relate to healthy eating behavior. Scoring for the TPB is the sum of each subscale. Attitude range of scores: 7-49 - higher score means greater/more positive attitude; SN range: 3-21 - higher score greater/more positive subjective norm; PBC range: 3-21 - higher score greater/more positive PBC; Intention range: 6-42 - higher score greater/more positive intention.
Self-Regulation Healthy Eating Constructs: Prospective/ Retrospective Control, Action Planning | Measured at pre-post intervention, daily during the 10-day free-living period, and weekly throughout the intervention study period (~6 months).
  Self-regulation of HE will be measured in order to inform our dynamical model and to how well OW/OBPW are at regulating their energy intake and expenditure and how it impacts their GWG.
  These items were taken from Ryan Rhodes items for self-regulation of PA and adapted for HE behaviors. Ryan has indicated that these items work really well as an index for HE self-regulation because these behaviors are naturally inter-connected but to look at specific self-regulatory behaviors: self-monitoring, goal-setting, action planning, coping planning, scheduling, affective There are also 2 sets of 8 questions-first 8 examine prospective behaviors while the second set assesses retrospective behaviors.
  Retrospective scores range from 11-55 and Prospective scores range from 11-55. Total scores range from 22-110. A higher score indicates higher levels of HE self-regulation.
Self-Regulation Physical Activity Constructs: Prospective/ Retrospective Control, Action Planning | Measured at pre-post intervention, daily during the 10-day free-living period, and weekly throughout the intervention study period (~6 months).
  Self-regulation of PA will be measured in order to inform our dynamical model and to how well OW/OBPW are at regulating their energy intake and expenditure and how it impacts their GWG. These items are taken from Ryan Rhodes. Ryan has indicated that these items work really well as an index because these behaviors are naturally inter-connected but to look at specific self-regulatory behaviors: Item #1: self-monitoring, Item #2: goal-setting, Item # 3: action planning, Item #4: coping planning, Item #5: scheduling, Item #6, 7, 8, 9: cuing, Items 10 & 11: affective. There are also 2 sets of 8 questions-first 8 examine prospective behaviors while the second set assesses retrospective behaviors. Retrospective scores range from 11-55 and Prospective scores range from 11-55. Total scores for overall self-regulation range from 22-110. A higher score indicates higher levels of PA self-regulation.
Resting Metabolic Rate | Measured at pre- and -post intervention of the 6 month intervention study period.
  RMR will be calculated using a quadratic regression formula. Our pilot data showed no significant difference and similar means in PW-OW/OB's RMR when it was measured with the Breezing mobile metabolism device vs. estimated with the equation, thus we will estimate RMR with the formula to reduce subject burden.
Diet Quality | Measured at pre-post intervention and weekly (3 days/week) throughout the intervention study period (~6 months).
  Self-reported diet quality will be assessed with the Smartphone app MyFitnessPal. Women will record their intake on at least 2 weekdays and 1 weekend per week over the study as a global indicator of their diet quality. This information will be used to personalize the intervention goals from week to week.
Pittsburgh Sleep Quality Index | Measured once at pre-post intervention and monthly throughout the intervention study period (~6 months)
  The Pittsburgh Sleep Quality Index (PSQI) is an 18-item valid/reliable measure to measure the quality and patterns of sleep in older adults. It differentiates "poor" from "good" sleep by measuring seven areas: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication and daytime dysfunction over the last month. The participant self-rates each of these seven areas of sleep. Scoring of answers is based on a 0 to 3 scale, whereby 3 reflects the negative extreme on the Likert Scale. Scores can range from 0-21. An overall sleep quality score greater than or equal to 5 reflects poor sleep quality. The outcome reported is overall sleep quality.
Sleep Behaviors - FitBit Charge 5 Activity Monitor | Measured daily at pre-post intervention and daily throughout the intervention study period (~6 months).
  The Fitbit Charge 5 will give a continuous PA measure in our energy balance model to predict GWG and assess sleep behaviors (time to sleep/wake, minutes of sleep/nighttime awakenings/light and deep rapid eye movement).
PROMIS Sleep Disturbance Short Form | Measured daily at pre-post intervention and daily throughout the study period (~6 months)
  The PROMIS Sleep Disturbance (PROMIS-SD) Short Form is an 8-item questionnaire that assesses sleep disturbances in individuals 18 or older. Each item rates the severity of the individual's sleep disturbance during the past 7 days. The measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of sleep disturbance.
Activity and Sleep Logs | Measured daily at pre-post intervention and daily throughout the study (~6 months)
  The PA log will track device use and monitor wear time (ActiGraph during pre-post intervention assessment period and Fitbit Charge 5 at pre- and post-intervention and throughout the study and the sleep log will also track time to bed and awake.
Three Factor Eating Questionnaire | Measured once at pre-post intervention and monthly throughout the intervention study period (~6 months)
  The Three Factor Eating Questionnaire is a 51-item questionnaire developed to measure three dimensions of human eating behavior: 1) dietary restraint, or cognitive control of eating behavior, 2) dietary disinhibition, or disinhibition of cognitive control of eating, and 3) susceptibility to hunger. The investigators are only using 18 items of the revised TFEQ. The TFEQ is examined by subscale scores and not by a total score. Subscale scores for the cognitive restraint scale range from 3-12; higher scores indicate higher levels of cognitive restraint of eating. Uncontrolled eating scale range from 9-36; higher scores indicate higher levels of uncontrolled eating behaviors. Emotional eating scale range from 6-24; higher scores indicate higher levels of emotional eating behaviors. Outcome measure results are reported as the score during the post-intervention week.
Infant Birth Outcomes | Measured at delivery of child. Data will be retrieved from medical records.
  Birth weight will be abstracted from the labor and delivery electronic health record along with infant length, sex, and gestational age and date of birth. These data will be used to determine infant birth weight for length based on percentiles for gestational age at delivery and sex estimated by the World Health Organization. In the event that birth weight data are missing or unavailable from the medical record, the investigators will obtain birth weight and related information from the participant's self-report.
Maternal-Infant Labor/Delivery and Adverse Pregnancy Outcomes | Measured at labor/delivery. Data will be retrieved from medical records.
  Labor and delivery data will be abstracted from the medical record and will include infant APGAR score, mode of delivery (vaginal or cesarean), and adverse pregnancy outcomes (e.g., diagnosis of gestational diabetes, insulin use, preeclampsia, depression, labor/delivery issues and other complications). In the event that labor/delivery data is missing or unavailable from the medical record, the investigators will obtain information from the participant's self-report.
Implementation Markers: Subject engagement/participation and acceptability | Through study completion, approximately 6 months
  Subject engagement/participation: fidelity monitoring will be conducted by a trained staff observer who will watch video recordings of 50% of intervention sessions and follow a review checklist to measure engagement (degree of subject responsiveness with session content, discussion, and activities.
  Subject acceptability: subjects and staff will be asked to complete weekly checklists to assess: attendance (0-100% attendance at pre/post-intervention sessions for all subjects; 0-100% attendance at baseline dosage/adaptive dosage sessions for intervention subjects); compliance (0-100% compliance with mHealth tools during free-living pre/post intervention sessions and daily [Wi-Fi weight scale, PA monitor], weekly [EI diet quality phone app, online surveys], and monthly [online surveys] for all subjects over the study period; 0-100% compliance with session activities); and quality/completeness of data (0-100% of usable data for each subject).
Implementation Markers: Subject Facilitators and Barriers | Measured at post-intervention, approximately at 34-37 weeks gestation
  N=12 women will be selected the interviews who had excellent compliance to get quality feedback on facilitators/benefits. N=13 women will be selected for interviews who had challenges with compliance to gain key insight about barriers. Interviews are expected to take 45-60 minutes.
Implementation Markers: Clinician Stakeholder Facilitators and Barriers | Measured at study completion and once all participants have completed the study, which could be roughly 2 years after start of study
  Feedback from key clinician stakeholders (i.e., registered dietitians, nurses, OB/Gyn providers; (N=20; n=10 HMC, n=10 Geisinger) will be obtained to understand facilitators/barriers to using the HMZ 2.0 digital platform. Clinicians will be asked to participate in a brief 10-min asynchronous training session that explains the HMZ 2.0 digital platform. They will then be asked to participate in a tutorial session using the HMZ web-based user interface to review an example patient's data, see graphical displays, manipulate PA/EI kcals to see correspondence with changes in predicted GWG, and review the host of recommended PA/EI strategies that will be recommended to implement with the patient. Semi-structured interviews with each clinician will be conducted to understand key facilitators/barriers to the platform.
Implementation Markers: Staff engagement, burden | Through study completion, approximately 6 months
  Staff engagement: fidelity monitoring will be conducted by a trained staff observer who will watch video recordings from the same sample of 50% of video recordings noted above and follow a review checklist to measure engagement (enthusiasm, preparedness, session delivery effectiveness, responsiveness to subject).
  Staff burden: weekly checklists completed by staff regarding amount of time spent preparing for sessions, responding to/following-up with subjects, using the HMZ 2.0 digital platform, and issues with delivering dosage recommendations to the subjects.
Implementation Markers: Dosage exposure | Through study completion, approximately 6 months
  Dosage exposure will be assessed by: a) weekly checklists completed by subjects/staff regarding amount of program content delivered/received (goal 90%+ coverage); b) fidelity monitoring by trained staff observer who will watch video recordings from the same sample of 50% of video recordings noted above; and c) tracking # of dosage changes determined by controller, # days between dosage change recommendation and implementation by staff, and type of active learning strategies in added dosages.

OTHER OUTCOMES:
Clinical/Safety Protocol: Height | Measured at pre-intervention
  Height will be assessed with a stadiometer using standard procedures in the Penn State Clinical Research Center.
Clinical/Safety Protocol: Blood Pressure/Urine | Measured at pre-intervention
  Blood pressure and urine BP>140/90, 1+ protein in urine) to will be measured/collected to (screen for preeclampsia at the Penn State Clinical Research Center.
Clinical/Safety Protocol: Socio-demographic Measures | Measured at pre-intervention
  Participants complete measures assessing general demographic information (e.g., age, pre-pregnancy BMI, race/ethnicity, marital status, family income, parity, medical history, smoking, drinking, other health-related behaviors, family health history, pregnancy history, and complications in any previous pregnancies they may have had that did go to full term.
Clinical/Safety Protocol: Center for Epidemiological Studies Depression Scale | Measured at pre-post intervention and monthly over the study for the safety protocol (~6 months)
  The Center for Epidemiological Studies Depression (CES-D) scale is a 20-item self-report scale that is designed to measure current levels of depressive symptomology (with emphasis on the affective component, depressed mood) in the general population. Scores can range from 0-60. A score of 16 or higher is indicative of depressive symptoms. Women with scores of 16 or higher will be referred for follow-up with their provider (or given a referral as needed).

CONTACTS AND LOCATIONS:
Locations (1):
- Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
To gain access to restricted data, researchers must submit a User Agreement and Distribution Agreement. The User Agreement specifies that the investigator will only use the data for the specific project as described. The User Agreement is not transferable to another recipient or facility and data may only be shared with others by obtaining them directly through the PI. The recipient must also agree to not attempt to establish the individual identities of participants who provided the data. The Distribution Agreement includes a detailed description of the proposed project. The proposal must include personal identification and institutional affiliation, a current resume, source of funding, a detailed summary of the proposed research including a statement of why publicly available data are insufficient, and a complete list of data requested, including data system, files, years, variables, and the like. The PI and a subcommittee of the research team will review all proposals.

REFERENCES:
- [Background] Gray NW, Fourgeaud L, Huang B, Chen J, Cao H, Oswald BJ, Hemar A, McNiven MA. Dynamin 3 is a component of the postsynapse, where it interacts with mGluR5 and Homer. Curr Biol. 2003 Mar 18;13(6):510-5. doi: 10.1016/s0960-9822(03)00136-2. PMID 12646135
- [Background] Garcia Compean D. [Treatment of acute hepatitis C]. Rev Gastroenterol Mex. 2002 Oct;67 Suppl 2:S61-6. Spanish. PMID 12712857
- [Background] Badon LA, Hicks A, Lord K, Ogden BA, Meleg-Smith S, Varner KJ. Changes in cardiovascular responsiveness and cardiotoxicity elicited during binge administration of Ecstasy. J Pharmacol Exp Ther. 2002 Sep;302(3):898-907. doi: 10.1124/jpet.302.3.898. PMID 12183645
- [Background] Calabresi L, Gomaraschi M, Villa B, Omoboni L, Dmitrieff C, Franceschini G. Elevated soluble cellular adhesion molecules in subjects with low HDL-cholesterol. Arterioscler Thromb Vasc Biol. 2002 Apr 1;22(4):656-61. doi: 10.1161/hq0402.105901. PMID 11950706
- [Derived] Khan O, Campregher F, Rivera DE, Visioli A, Pauley AM, Downs DS. An Optimized Behavioral Intervention for Managing Gestational Weight Gain Using Semi-Physical Modeling and Hybrid Model Predictive Control. IEEE Int Conf Commun. 2025 Jul;2025:3317-3322. doi: 10.23919/ACC63710.2025.11107916. Epub 2025 Aug 21. PMID 41306560